CLINICAL TRIAL: NCT02097238
Title: A Phase II Study of Eribulin (NSC# 707389) in Recurrent or Refractory Osteosarcoma
Brief Title: Eribulin Mesylate in Treating Patients With Recurrent or Refractory Osteosarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2014-00621; NCI-2014-00621 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); COG-AOST1322; AOST1322 (Other: Children's Oncology Group); AOST1322 (Other: CTEP); U10CA180886 (NIH); U10CA098543 (NIH)
Record Dates: First submitted 2014-03-24; First posted 2014-03-27 (Estimated); Results first posted 2017-09-01 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Recurrent Osteosarcoma
MeSH Terms: conditions — Osteosarcoma | interventions — eribulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (eribulin mesylate) (Experimental): Patients receive eribulin mesylate IV over 2-5 minutes on days 1 and 8. Courses repeat every 21 days for up to 24 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Eribulin Mesylate; Other: Pharmacological Study

INTERVENTIONS:
Drug: Eribulin Mesylate — Given IV
  Other Names: E7389; ER-086526; Halaven; Halichondrin B Analog
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase II trial studies how well eribulin mesylate works in treating patients with osteosarcoma that has come back after treatment (recurrent) or has not responded to treatment (refractory). Microtubule inhibitors, such as eribulin mesylate, may stop or slow the growth of tumor cells by disrupting the cell cycle.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the 4 month progression free survival rate and objective response rate in patients with recurrent osteosarcoma who are administered eribulin (eribulin mesylate) therapy on day 1 and day 8 of 21 day cycles.

SECONDARY OBJECTIVES:

I. To investigate the pharmacokinetics (PK) of eribulin in subjects with recurrent osteosarcoma.

II. To further describe the tolerability of single agent eribulin.

OUTLINE:

Patients receive eribulin mesylate intravenously (IV) over 2-5 minutes on days 1 and 8. Courses repeat every 21 days for up to 24 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up annually for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have had histologic verification of osteosarcoma at original diagnosis
* Patients must have measurable disease, documented by clinical, radiographic, or histologic criteria, and have relapsed or become refractory to conventional therapy
* Patients must have a performance status corresponding to Eastern Cooperative Oncology Group (ECOG) scores of 0, 1 or 2; use Karnofsky for patients > 16 years of age and Lansky for patients =< 16 years of age
* Patients must have a life expectancy of >= 8 weeks
* Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study

  * Myelosuppressive chemotherapy: must not have received within 2 weeks of entry onto this study (6 weeks if prior nitrosourea)
  * Biologic (anti-neoplastic agent): at least 7 days since the completion of therapy with a biologic agent
  * Bisphosphonates: at least 4 weeks since the completion of therapy with a bisphosphonate
  * Monoclonal antibodies: at least 3 half-lives must have elapsed since prior therapy that included a monoclonal antibody
  * Radiation therapy (RT): >= 2 weeks (wks) for local palliative RT (small port); >= 6 months must have elapsed if prior craniospinal RT or if >= 50% radiation of pelvis; >= 6 weeks must have elapsed if other substantial bone marrow (BM) radiation
* Peripheral absolute neutrophil count (ANC) >= 1000/uL
* Platelet count >= 75,000/uL (transfusion independent)
* Hemoglobin >= 8.0 g/dL (may receive red blood cell [RBC] transfusions)
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^2 or
* A serum creatinine based on age/gender as follows: (threshold creatinine values were derived from the Schwartz formula for estimating GFR)

  * Age (12 to < 13 years) - serum creatinine of 1.2 mg/dL
  * Age (13 to < 16 years) - serum creatinine of 1.5 mg/dL (male) and 1.4 mg/dL (female)
  * Age (>= 16 years) - serum creatinine of 1.7 mg/dL (male) and 1.4 mg/dL (female)
* Bilirubin (sum of conjugate + unconjugated) =< 1.5 x upper limit of normal (ULN) for age
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 110 units per liter (U/L); for the purpose of this study, the ULN for SGPT is 45 U/L
* Serum albumin > 2 g/dL
* Shortening fraction of >= 27% by echocardiogram
* Ejection fraction of >= 50% by radionuclide angiogram
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Exclusion Criteria:

* Patients with congenital prolonged QT syndrome
* Patients with a baseline QT/corrected QT (QTc) interval >= 501 msec
* Patients who are receiving drugs that prolong the QTc are not eligible
* Patients who have previously received eribulin, halichondrin B, or analogues of halichondrin B
* Patients who have grade >= 2 peripheral neuropathy
* Patients who are receiving other cancer directed therapy at the time of enrollment
* Patients who have had major surgery within 3 weeks prior to enrollment are not eligible; procedures such as placement of a central vascular catheter, or limited tumor biopsy, are not considered major surgery
* Pregnancy and breast feeding

  * Female patients who are pregnant are ineligible
  * Lactating females are not eligible unless they have agreed not to breastfeed their infants
  * Female patients of childbearing potential are not eligible unless a negative pregnancy test result has been obtained
  * Sexually active patients of reproductive potential are not eligible unless they have agreed to use an effective contraceptive method for the duration of their study participation

Ages: 12 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2020-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Isakoff, Principal Investigator — Children's Oncology Group
Locations (119):
- United States (116):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Southern California Permanente Medical Group, Downey, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Mattel Children's Hospital UCLA, Los Angeles, California
  - Children's Hospital Central California, Madera, California
  - Children's Hospital and Research Center at Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Hospital, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Memorial University Medical Center, Savannah, Georgia
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Maine Children's Cancer Program, Scarborough, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Michigan State University Clinical Center, East Lansing, Michigan
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Medical Center-Fairview, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Central Care Cancer Center-Carrie J Babb Cancer Center, Bolivar, Missouri
  - CoxHealth Cancer Center, Branson, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital-Joplin, Joplin, Missouri
  - The Childrens Mercy Hospital, Kansas City, Missouri
  - Phelps County Regional Medical Center, Rolla, Missouri
  - Saint John's Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - 21st Century Oncology - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - 21st Century Oncology, Las Vegas, Nevada
  - Children's Specialty Center of Nevada II, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - 21st Century Oncology - Fort Apache, Las Vegas, Nevada
  - Cancer and Blood Specialists-Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - 21st Century Oncology - Vegas Tenaya, Las Vegas, Nevada
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Columbia University Medical Center, New York, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Mission Hospital-Memorial Campus, Asheville, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Sanford Medical Center-Fargo, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - The Toledo Hospital/Toledo Children's Hospital, Toledo, Ohio
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Palmetto Health Richland, Columbia, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Childrens Hospital-King's Daughters, Norfolk, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
- Canada (3):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Eribulin Mesylate)
Started | 19
Completed | 0
Not Completed | 19
Not completed — Death | 1
Not completed — Physician Decision | 1
Not completed — Progressive Disease | 17

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Eribulin Mesylate)
Number analyzed (Participants) | 19
Age, Continuous [Mean (Full Range); unit: Years] | 17 [12 to 25]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 14
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: Participants]
  Canada | 2
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Disease Control Success
Description: The number of patients who do not experience disease progression or death in the four months following enrollment on AOST1322.
Time Frame: 4 Months
Measure: Number; unit: participants
Arm/Group | Treatment (Eribulin Mesylate)
Number analyzed (Participants) | 19
participants | 0

2. Primary Outcome: Response Evaluation Criteria in Solid Tumors (RECIST) Response
Description: The number of patients who experience a complete or partial response according to the RECIST criteria as defined in Eisenhauer et al. Eur J Cancer 45:228-47, 2009.
Time Frame: 4 months
Measure: Number; unit: participants
Arm/Group | Treatment (Eribulin Mesylate)
Number analyzed (Participants) | 19
participants | 0

3. Secondary Outcome: Number of Cycles Where a Dose Limiting Toxicity Was Identified
Description: Each cycle where the patient receives eribulin and does not receive non-protocol anticancer therapy will be considered in the analysis. A dose limiting toxicity is defined to be: day 8 eribulin dose is held due to grade 3 or grade 4 non-hematological toxicity attributable to the investigational drug and does not resolve to meet eligibility or baseline criteria by day 11. Any >= grade 3 non-hematological toxicity attributable to the investigational drug with the specific exclusion of: grade 3 nausea and vomiting < 3 days duration grade 3 liver enzyme elevation, including alanine aminotransferase (ALT)/aspartate aminotransferase (AST)/gamma-glutamyltransferase (GGT), that returns to grade =< 1 or baseline prior to the time for the next treatment cycle.
Time Frame: 4 months
Population: 19 patients were treated on protocol therapy. Thirty-nine cycles were reported for the analysis of dose limiting toxicity.
Measure: Number; unit: Cycles
Units Other Than Participants: Cycles
Arm/Group | Treatment (Eribulin Mesylate)
Number analyzed (Participants) | 19
Number analyzed (Cycles) | 39
Cycles | 2

4. Secondary Outcome: Area Under the Curve 0-infinity of Eribulin Mesylate in Ng-hr/ml
Description: Data from all patients who provide samples for pharmacokinetic analysis will be aggregated. The sample mean and variance of the area under the curve will be reported The analytic unit will be the patient-cycle: Each cycle where the patient receives eribulin and does not receive non-protocol anticancer therapy will be considered in the analysis.
Time Frame: Cycle 1 day 1 and cycle 2 day 1 at the end of infusion, 0.5-6 hours, and 24-120 hours post infusion; cycle 1 day 8 and cycle 2 day 8 prior to the dose of eribulin and at the end of infusion
Population: 5 patients contributed 9 cycles for the calculation of the sample mean and standard deviation of Area under the curve
Measure: Mean (Standard Deviation); unit: hour-nanograms/mL
Units Other Than Participants: patient-cycles
Arm/Group | Treatment (Eribulin Mesylate)
Number analyzed (Participants) | 5
Number analyzed (patient-cycles) | 9
hour-nanograms/mL | 2475.293034 (1746.75558)

5. Secondary Outcome: Clearance of Eribulin Mesylate in L/hr
Description: Data from all patients who provide samples for pharmacokinetic analysis will be aggregated. The sample mean and variance of the clearance will be reported. The analytic unit will be the patient-cycle: Each cycle where the patient receives eribulin and does not receive non-protocol anticancer therapy will be considered in the analysis.
Time Frame: as for outcome 4
Population: 5 patients contributed 9 cycles for the calculation of the sample mean and standard deviation of clearance
Measure: Mean (Standard Deviation); unit: L/hour
Units Other Than Participants: patient-cycles
Arm/Group | Treatment (Eribulin Mesylate)
Number analyzed (Participants) | 5
Number analyzed (patient-cycles) | 9
L/hour | 1.585078903 (1.08079608)

6. Secondary Outcome: A Half Life of Eribulin Mesylate in hr
Description: Data from all patients who provide samples for pharmacokinetic analysis will be aggregated. The sample mean and variance of the half life will be reported. The analytic unit will be the patient-cycle: Each cycle where the patient receives eribulin and does not receive non-protocol anticancer therapy will be considered in the analysis.
Time Frame: 1 day 1 and cycle 2 day 1 at the end of infusion, 0.5-6 hours, and 24-120 hours post infusion; cycle 1 day 8 and cycle 2 day 8 prior to the dose of eribulin and at the end of infusion
Population: 5 patients contributed 9 cycles for the calculation of the sample mean and standard deviation of half life
Measure: Mean (Standard Deviation); unit: hours
Units Other Than Participants: patient-cycles
Arm/Group | Treatment (Eribulin Mesylate)
Number analyzed (Participants) | 5
Number analyzed (patient-cycles) | 9
hours | 40.22202016 (2475.293034)

ADVERSE EVENTS:
Arm/Group | Treatment (Eribulin Mesylate)
Serious Adverse Events (participants affected / at risk) | 10/19
Other Adverse Events (participants affected / at risk) | 6/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Eribulin Mesylate) (N=19)
Pericardial effusion (Cardiac disorders) | 1 (1)
Papilledema (Eye disorders) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Eribulin Mesylate) (N=19)
Neutrophil count decreased (Investigations) | 4 (4)
White blood cell decreased (Investigations) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less